CLINICAL TRIAL: NCT04951206
Title: A Randomized Controlled Trial of Vulvar Fractionated CO2-Laser Therapy With and Without Concomitant Topical Clobetasol Propionate 0.05% Ointment for Treatment of Vulvar Lichen Sclerosus
Brief Title: Fractionated CO2 Laser With and Without Clobetasol for Treatment of Vulvar Lichen Sclerosus
Acronym: VULVIE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Patty Brisben Foundation For Women's Sexual Health (Other); Society of Gynecologic Surgeons (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHRI IRB #STUDY00003851
Record Dates: First submitted 2021-06-22; First posted 2021-07-06 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Vulvar Lichen Sclerosus
Keywords: Clobetasol propionate; Fractionated CO2-laser
MeSH Terms: conditions — Vulvar Lichen Sclerosus | interventions — Clobetasol; Ointments

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clobetasol Group (Active Comparator): Clobetasol propionate 0.05% ointment is the active treatment arm that will be use in women with lichen sclerosus in the study per standard clinical recommendations. Participants will be instructed to apply 0.25-0.5g of the ointment to the affected tissues nightly for 4 weeks starting after the initial FxCO2 laser treatment, then 2 times a week for the remainder of the study (until final study visit).
  Interventions: Device: Fractionated CO2-laser; Drug: Clobetasol Propionate 0.05% Ointment
- Placebo Group (Placebo Comparator): Placebo ointment is the control treatment arm. Participants will be instructed to apply 0.25-0.5g of the ointment to the affected tissues nightly for 4 weeks starting after the initial FxCO2 laser treatment, then 2 times a week for the remainder of the study (until final study visit).
  Interventions: Device: Fractionated CO2-laser

INTERVENTIONS:
Device: Fractionated CO2-laser — All women will be undergoing FxCO2-laser therapy as this treatment is a criterion for enrollment.
Drug: Clobetasol Propionate 0.05% Ointment — Clobetasol propionate 0.05% ointment obtained from a commercial manufacturer
  Other Names: Clobetasol
  Arms: Clobetasol Group

SUMMARY:
This is a randomized placebo-controlled trial design to determine whether combining FxCO2-laser with the traditional therapy of clobetasol propionate 0.05% ointment (combined treatment) as compared to FxCO2-laser and placebo ointment (FxCO2-laser only) will improve treatment response in women undergoing FxCO2-laser for vulvar lichen sclerosus.

Primary objective: To evaluate if women with LS who undergo FxCO2 laser therapy and concomitant TCS (clobetasol group) have higher treatment success (defined as a MCID of a ≥16 point improvement in Skindex-29 questionnaire) than those who undergo FxCO2 laser and placebo ointment (placebo group).

* Hypothesis: A higher proportion of women randomized to clobetasol will achieve treatment success as compared to those randomized to placebo.
* Approach: The proportion of women in each cohort who obtain a ≥16 point improvement in Skindex-29 validated questionnaire score from baseline to final visit will be compared.

Secondary objectives: To compare change in pre- and post-treatment scores on validated questionnaires measuring vulvovaginal symptoms, sexual function, lower urinary tract function, and genital self-image between the clobetasol group compared to the placebo group.

* Hypothesis: Women randomized to clobetasol will demonstrate an equal or greater improvement on validated quality of life questionnaires measuring vulvovaginal symptoms, sexual function, lower urinary tract function, and genital self-image as compared to women randomized to placebo.
* Approach: Change scores will be calculated to determine change per participant over the treatment period and mean change scores will be compared between cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years old with biopsy confirmed or clinically diagnosed+ LS
* English-speaking or Spanish-speaking
* Electing to undergo Fractionated CO2-laser therapy
* Willing and able to undergo concomitant 0.05% clobetasol propionate treatment

Exclusion Criteria:

* Prior surgery with placement vaginal mesh for repair of pelvic organ prolapse (does not include vaginal mesh for anti-incontinence procedure "sling" or prior mesh sacrocolpopexy)
* Prior laser, topical immunomodulators or systemic therapy for LS
* Active genital infection^
* Suspicious vulvar lesion that has not been evaluated
* Known vulvar or vaginal malignancy or active treatment for other malignancy
* Planning pregnancy or pregnant
* Prior pelvic radiation therapy
* Topical corticosteroid use on the vulvovaginal tissues in the past 2 weeks*
* Contraindication or allergy to clobetasol propionate 0.05%
* Currently breast-feeding or lactating
* History of poor wound healing, keloids or hypertrophic scarring
* History of a skin condition that could interfere with evaluation of efficacy and safety

  * Eligible for inclusion after washout period of 2 weeks ^Eligible for inclusion after treatment. For patients with known genital HSV we will instruct them to remain on suppression for the duration of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is investigating treatment of vulvar lichen sclerosus and thus participants will be limited to women with vulvar lichen sclerosus
Enrollment: 212 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-04-25 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Treatment success | About 5 months (baseline to final visit)
  Minimally clinically important difference of a ≥16 point improvement in Skindex-29 validated questionnaire score. Skindex-29 responses are transformed to a linear scale from 0 (no effect) to 100 (effect experienced all the time), and are reported as three scale scores, corresponding to three domains (symptoms, emotions, and functioning). A reduction in Skindex-29 score of 16 points or more has been shown to indicate what is considered a clinically meaningful improvement.

SECONDARY OUTCOMES:
Treatment response - vulvovaginal symptoms | About 5 months (baseline to final visit)
  Treatment response - vulvovaginal symptoms will be measured by pre- and post-treatment scores on the vulvovaginal Symptoms Questionnaire, a 21-item survey measuring vulvovaginal symptoms in postmenopausal women.
Treatment response - sexual function | About 5 months (baseline to final visit)
  Treatment response - sexual function will be measured by pre- and post-treatment scores on the Female Sexual Function Index, a validated questionnaire to assess sexual function.
Treatment response - genital self image | About 5 months (baseline to final visit)
  Treatment response - genital self image will be measured by pre- and post-treatment scores on the Female Genital Self Image Scale, a validated survey with scores ranging from 7-28 with higher scores indicate a more positive genital self-image.
Treatment response - lower urinary tract function | About 5 months (baseline to final visit)
  Treatment response - lower urinary tract function will be measured by pre- and post-treatment scores on the LURN SI-10, a 10-item questionnaire with scores ranging from 0 to 38 (higher scores = worse symptoms/bother).
Participant-perceived improvement | Final study visit at 4-6 weeks after third Fractionated CO2 laser treatment - one time question
  Patient Global Impression of Improvement (PGI-I): a one single item question that will ask participants to rate their improvement after undergoing treatment on a 7-point Likert scale ranging from "very much worse" to "very much better."
Participant-perceived treatment satisfaction | Final study visit at 4-6 weeks after third Fractionated CO2 laser treatment - one time question
  Level of satisfaction with treatment: a one single item question that will ask participants to rate their level of satisfaction with treatment on a 5-point Likert scale from "very dissatisfied" to "very satisfied".

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Kaiser Permanente - Southern California Permanente Medical Group, San Diego, California
  - MedStar Health, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - The University of New Mexico, Albuquerque, New Mexico
  - Columbia University, New York, New York
  - Ohio State University, Columbus, Ohio
  - The Institute for Female Pelvic Medicine & Reconstructive Surgery, Allentown, Pennsylvania
  - Waukesha Memorial Hospital, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chren MM. The Skindex instruments to measure the effects of skin disease on quality of life. Dermatol Clin. 2012 Apr;30(2):231-6, xiii. doi: 10.1016/j.det.2011.11.003. Epub 2011 Dec 20. PMID 22284137
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Herbenick D, Schick V, Reece M, Sanders S, Dodge B, Fortenberry JD. The Female Genital Self-Image Scale (FGSIS): results from a nationally representative probability sample of women in the United States. J Sex Med. 2011 Jan;8(1):158-66. doi: 10.1111/j.1743-6109.2010.02071.x. Epub 2010 Nov 2. PMID 21044269
- [Background] Herbenick D, Reece M. Development and validation of the female genital self-image scale. J Sex Med. 2010 May;7(5):1822-30. doi: 10.1111/j.1743-6109.2010.01728.x. Epub 2010 Mar 3. PMID 20233278
- [Background] Hodges KR, Wiener CE, Vyas AS, Turrentine MA. The Female Genital Self-image Scale in Adult Women With Vulvar Lichen Sclerosus. J Low Genit Tract Dis. 2019 Jul;23(3):210-213. doi: 10.1097/LGT.0000000000000481. PMID 31135654
- [Background] Cella D, Smith AR, Griffith JW, Kirkali Z, Flynn KE, Bradley CS, Jelovsek JE, Gillespie BW, Helfand BT, Talaty P, Weinfurt KP; LURN Study Group. A New Brief Clinical Assessment of Lower Urinary Tract Symptoms for Women and Men: LURN SI-10. J Urol. 2020 Jan;203(1):164-170. doi: 10.1097/JU.0000000000000465. Epub 2019 Jul 31. PMID 31364922
- [Background] Erekson EA, Yip SO, Wedderburn TS, Martin DK, Li FY, Choi JN, Kenton KS, Fried TR. The Vulvovaginal Symptoms Questionnaire: a questionnaire for measuring vulvovaginal symptoms in postmenopausal women. Menopause. 2013 Sep;20(9):973-9. doi: 10.1097/GME.0b013e318282600b. PMID 23481118